CLINICAL TRIAL: NCT03782363
Title: A Phase I Study of Adoptive Immunotherapy With Cytokine-Induced Killer Cells in Relapsed and Non-resectable Sarcomas After Multimodal Treatment.
Brief Title: Study of Adoptive Immunotherapy in Relapsed and Non-resectable Sarcomas After Multimodal Treatment.
Acronym: CAST
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Initial version of the protocol not submitted and new version approved has a new sponsor and it has been added into Clinicaltrials by the new sponsor
Sponsor: Italian Sarcoma Group (Network)
Collaborators: Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ISG-CAST
Record Dates: First submitted 2018-12-17; First posted 2018-12-20 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Sarcoma
Keywords: advanced sarcoma; osteosarcoma; soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma

STUDY DESIGN:
Intervention Model Description: Dose finding study for the determination of the MTD for the RP2D with cohort of 3 patients plus 3 other patients as scaling design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Autologous CIK Dose level 1 (Experimental): autologous CIK at dose level 1
  Interventions: Biological: Autologous CIK Dose level 1
- Autologous CIK Dose level 2 (Experimental): autologous CIK at dose level 2
  Interventions: Biological: Autologous CIK Dose level 2
- Autologous CIK Dose level 3 (Experimental): autologous CIK at dose level 3
  Interventions: Biological: Autologous CIK Dose level 3
- Autologous CIK Dose level 4 (Experimental): autologous CIK at dose level 4
  Interventions: Biological: Autologous CIK Dose level 4

INTERVENTIONS:
Biological: Autologous CIK Dose level 1 — Lymphocytapheresis of the autologous ex-vivo CIK cell expanded in the Cell factory at first level of dose 20.000.000 cell/kgs days 1 and 22
  Arms: Autologous CIK Dose level 1
Biological: Autologous CIK Dose level 2 — Lymphocytapheresis of the autologous ex-vivo CIK cell expanded in the Cell factory at first level of dose 25.000.000 cell/kgs days 1 and 22
  Arms: Autologous CIK Dose level 2
Biological: Autologous CIK Dose level 3 — Lymphocytapheresis of the autologous ex-vivo CIK cell expanded in the Cell factory at first level of dose 20.000.000 cell/kgs days 1 and 15
  Arms: Autologous CIK Dose level 3
Biological: Autologous CIK Dose level 4 — Lymphocytapheresis of the autologous ex-vivo CIK cell expanded in the Cell factory at first level of dose 25.000.000 cell/kgs days 1 and 15
  Arms: Autologous CIK Dose level 4

SUMMARY:
Monocentric, phase I study for advanced sarcoma with adoptive immunotherapy with Cytokine-Induced Killer (CIK).

In the first part of the study Patient's' peripheral blood will be collected and CIK cell expansion and storage will occur at the Regina Margherita Children's Hospital Cell Factory.

In the second part of the study the Maximum Tolerated Dose (MTD) will be determined in order to find the Recommended Dose for Phase II (RP2D)

DETAILED DESCRIPTION:
In the first part of the study the patient's' peripheral blood collected from and CIK cell expansion and storage at the Regina Margherita Children's Hospital Cell Factory.

Approximately 40 patients will be enrolled in part 1 (range: 30 - 50 patients). The second part of the study will be a 3+3 dose escalation design to determine the MTD/RP2D.

A Safety Monitoring Committee (SMC) will be appointed to make dose escalation decisions.

Approximately 30 patients will be enrolled in this part (range: 6 - 36 patients).

Only one infusion of autologous CIK cells will be carried out at each cycle, every 21 days at the 1st, 2nd and 3rd dose levels and every 15 days at the 4th, 5th 6th dose levels.

A maximum of 6 cycles will be performed (patient with complete disease remission patients who benefit from treatment might also receive more cycles at the Investigator's discretion)

ELIGIBILITY:
Inclusion Criteria for part 1

1. Patients with histologically documented unresectable sarcomas which progressed after first or further line treatments for relapsing disease who could be enrolled in Part 2 of study immediately or after a new line of treatment;
2. Karnofsky score ≥ 70% (patients with Karnofsky score ≥ 50% are eligible if it depends solely on orthopedic problems)
3. Estimated life expectancy > 3 months;
4. Adequate bone marrow functions:
5. Signed informed consent;
6. Negative serum or urine pregnancy test within 48 hours from collection of peripheral blood or from lympho cyto apheresis (if post-pubertal female patients);
7. Archived histological tumour sample available

Inclusion Criteria for part 2

1. Patients with histologically documented unresectable sarcomas which progressed after a first or further line treatments for relapsing disease
2. Measurable disease (bone lesions are included);
3. Karnofsky score ≥ 70% (patients with Karnofsky score ≥ 50% are eligible if its depend solely on orthopedic problems)
4. Estimated life expectancy > 3 months;
5. Adequate bone marrow, hepatic and renal functionality
6. Signed informed consent;
7. Archived histological tumour sample available;
8. Patients should have a venous central access;
9. Pregnancy test should be negative 48 hours before treatment for post-pubertal women patients. All post-pubertal patients are to take adequate anti-contraceptive measures during treatment and until 8 weeks after the last dose of treatment.

Exclusion Criteria for part 1

1. History of Human Immunodeficiency Virus, Hepatitis C Virus, Hepatitis B Virus or Hepatitis A Virus infection;
2. Patients receiving chemotherapy and/or immunotherapy and/or anti-tumour agents and/or radiotherapy on more than 10% of bone marrow area two weeks before peripheral blood collection or lymphocytapheresis;
3. Patients with neuro-psychiatric disorders or social or geographic problems that would prohibit the understanding or rendering informed consent and compliance with the requirements of this protocol are excluded.

Exclusion Criteria for part 2

1. Patients with Ewing/Primitive Neuroectodermal Tumor Sarcoma, Rhabdomyosarcoma as well as other rapidly growing sarcomas are not to be included in the study;
2. Presence of Central Nervous System metastases and/or meningeal neoplastic involvement;
3. Patients with seizure disorders;
4. Severe renal, vascular, cardiac, hepatic, lung disorders;
5. Patients with any severe and/or uncontrolled medical conditions such as unstable angina pectoris, heart failure ≥ grade 2, a recent heart attack within 6 months, uncontrolled heart non arrhythmia uncontrolled metabolic disorders, cirrhosis, uncontrolled hypertension
6. Patients with a non-optimal ex-vivo expansion of autologous CIK cells during Part 1 (< 0.5 x 107/kg CIK cells);
7. History of Human Immunodeficiency Virus, Hepatitis C Virus, Hepatitis B Virus or Hepatitis A Virus infection;
8. Presence of bleeding disorders;
9. Patients undergoing renal dialysis;
10. Presence of uncontrolled diabetes
11. Patients unable to swallow oral medications;
12. Patients receiving concomitant steroid or immunotherapy (except corticosteroids with a daily dosage equivalent to prednisone ≤ 20 mg for adrenal insufficiency).
13. Anticancer chemotherapy or experimental drugs or immunotherapy or radiotherapy 2 weeks before entering the study;
14. Anticancer chemotherapy or experimental drugs or immunotherapy or radiotherapy on target lesions 2 weeks before entering the study;
15. Prior exposure to CIK cells;
16. Major surgery 4 weeks before entering the study;
17. Minor surgery 1 week before entering the study;
18. Patients with allergic reactions or hypersensibility to excipient
19. Pregnant or breast-feeding patients;
20. Patients with neuro-psychiatric disorders or social or geographic problems that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol are excluded.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) associated with CIK autologous cells administration | at week 6
  The MTD will be determined through dose-escalation using a 3+3 cohort design. If less than oner third of evaluable patients in a given cohort (0 of 3 patients or 1 of 6 patients) experiences a DLT; escalation may proceed to the next higher dose level.
  If one of the first 3 patients enrolled in a given cohort experiences a DLT, at least 3 additional patents will be enrolled in that cohort.
  If a DLT is observed in one-third or more of patients, the dose at which this occurs will be considered not tolerated and the MTD will have been exceeded. The highest dose level(s) at which less than one-third of patients (0 of 3 patients or 1 of 6 patients) experiences a DLT will be declared the MTD and will be used as RP2D

SECONDARY OUTCOMES:
Plasma concentration of autologous CIK cells for pharmacokinetic | At every cycle up to cycle 6 at: a) day 1 pre-dose b) 4 hours post-infusion, c) 24 hours post-infusion, d) day8 , e) day 15
  Evaluation of the plasma concentration of autologous CIK cells to determine the pharmacokinetics parameter of the autologous CIK cells
Progression free Survival | At month 4
  Survival free of disease progression
Evaluation of Major histocompatibility complex class I-related chains A and B on tumor material | pre-dose
  Major histocompatibility complex class I-related chains A and B expression in the tumor
Evaluation of UL16 binding proteins on tumor material | pre-dose
  UL16 binding proteins expression in the tumor
Quality of live reported by the Patients Using European Organisation of Research and Treatment (EORTC) Quality of Life Questionnaire Questionnaire-Core 30 (QLQ-C30) | at week 6
  Evaluation of the quality of life during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Franca Faggioli, MD, Principal Investigator — Ospedale Infantile Regina Margherita - Unit of Paediatric Oncoematology
Locations (1):
- Ospedale Infantile Regina Margherita - Unit of Paediatric Oncoematology, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt-Wolf IG, Lefterova P, Mehta BA, Fernandez LP, Huhn D, Blume KG, Weissman IL, Negrin RS. Phenotypic characterization and identification of effector cells involved in tumor cell recognition of cytokine-induced killer cells. Exp Hematol. 1993 Dec;21(13):1673-9. PMID 7694868
- [Background] Introna M, Franceschetti M, Ciocca A, Borleri G, Conti E, Golay J, Rambaldi A. Rapid and massive expansion of cord blood-derived cytokine-induced killer cells: an innovative proposal for the treatment of leukemia relapse after cord blood transplantation. Bone Marrow Transplant. 2006 Nov;38(9):621-7. doi: 10.1038/sj.bmt.1705503. Epub 2006 Sep 18. PMID 16980990
- [Background] Mesiano G, Todorovic M, Gammaitoni L, Leuci V, Giraudo Diego L, Carnevale-Schianca F, Fagioli F, Piacibello W, Aglietta M, Sangiolo D. Cytokine-induced killer (CIK) cells as feasible and effective adoptive immunotherapy for the treatment of solid tumors. Expert Opin Biol Ther. 2012 Jun;12(6):673-84. doi: 10.1517/14712598.2012.675323. Epub 2012 Apr 14. PMID 22500889
- [Background] Olioso P, Giancola R, Di Riti M, Contento A, Accorsi P, Iacone A. Immunotherapy with cytokine induced killer cells in solid and hematopoietic tumours: a pilot clinical trial. Hematol Oncol. 2009 Sep;27(3):130-9. doi: 10.1002/hon.886. PMID 19294626
- [Background] Heimann TG, Githens S. Rat pancreatic duct epithelium cultured on a porous support coated with extracellular matrix. Pancreas. 1991 Sep;6(5):514-21. doi: 10.1097/00006676-199109000-00003. PMID 1946307
- [Background] Gammaitoni L, Giraudo L, Macagno M, Leuci V, Mesiano G, Rotolo R, Sassi F, Sanlorenzo M, Zaccagna A, Pisacane A, Senetta R, Cangemi M, Cattaneo G, Martin V, Coha V, Gallo S, Pignochino Y, Sapino A, Grignani G, Carnevale-Schianca F, Aglietta M, Sangiolo D. Cytokine-Induced Killer Cells Kill Chemo-surviving Melanoma Cancer Stem Cells. Clin Cancer Res. 2017 May 1;23(9):2277-2288. doi: 10.1158/1078-0432.CCR-16-1524. Epub 2016 Nov 4. PMID 27815354
- [Background] Chan JK, Hamilton CA, Cheung MK, Karimi M, Baker J, Gall JM, Schulz S, Thorne SH, Teng NN, Contag CH, Lum LG, Negrin RS. Enhanced killing of primary ovarian cancer by retargeting autologous cytokine-induced killer cells with bispecific antibodies: a preclinical study. Clin Cancer Res. 2006 Mar 15;12(6):1859-67. doi: 10.1158/1078-0432.CCR-05-2019. PMID 16551871
- [Background] Kim HM, Lim J, Yoon YD, Ahn JM, Kang JS, Lee K, Park SK, Jeong YJ, Kim JM, Han G, Yang KH, Kim YJ, Kim Y, Han SB. Anti-tumor activity of ex vivo expanded cytokine-induced killer cells against human hepatocellular carcinoma. Int Immunopharmacol. 2007 Dec 15;7(13):1793-801. doi: 10.1016/j.intimp.2007.08.007. Epub 2007 Aug 31. PMID 17996690
- [Background] Schmidt-Wolf IG, Finke S, Trojaneck B, Denkena A, Lefterova P, Schwella N, Heuft HG, Prange G, Korte M, Takeya M, Dorbic T, Neubauer A, Wittig B, Huhn D. Phase I clinical study applying autologous immunological effector cells transfected with the interleukin-2 gene in patients with metastatic renal cancer, colorectal cancer and lymphoma. Br J Cancer. 1999 Nov;81(6):1009-16. doi: 10.1038/sj.bjc.6690800. PMID 10576658